CLINICAL TRIAL: NCT05960370
Title: Impact of Endometrial Compaction on Reproductive Outcomes After Cryotransfer of Euploid Embryos in a Natural Cycle: Prospective Cohort Study
Brief Title: Impact of Endometrial Compaction on Reproductive Outcomes After Cryotransfer of Euploid Embryos in a Natural Cycle
Acronym: Compaction
Status: Recruiting | Type: Observational
Sponsor: Instituto Bernabeu (Other)
Collaborators: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, Dr. Esperanza de la Torre Perez, Gynecologist, Instituto Bernabeu
Other Study IDs: Compaction Study
Record Dates: First submitted 2023-07-17; First posted 2023-07-25 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Infertility Due to Nonimplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- exposed or "compaction" group: 103 women with a decrease of ≥ 5% in endometrial thickness between the estrogenic phase (ovulation induction day) and the day of embryo transfer (7 days after ovulation induction).
  Interventions: Other: Observational non intervention study
- non-exposed "non-compaction" group: 103 women with similar or greater endometrial thickness between the estrogenic phase (ovulation induction day) and the day of embryo transfer (7 days after ovulation induction).
  Interventions: Other: Observational non intervention study

INTERVENTIONS:
Other: Observational non intervention study — An additional control scan will be performed vaginally the day of the embryo transfer. Rest of follow up and treatment will be executed as usually.

SUMMARY:
Multicenter prospective observational cohort study, comparing ongoing pregnancy rates in natural cycles for euploid embryo transfer in patients who present endometrial compaction at the time of the transfer versus those who have a stable or greater endometrial thickness with respect to the estrogenic phase.

DETAILED DESCRIPTION:
Multicenter prospective observational cohort study. Based on our sample size calculation, the study group will consist of 206 women (exposed or "compaction" group: 103 women with a decrease of ≥ 5% in endometrial thickness between the estrogenic phase and the day of embryo transfer; non-exposed "non-compaction" group: 103 women with similar or greater endometrial thickness between these time points). The main objective of this study is to compare the ongoing pregnancy rates in natural cycles for euploid embryo transfer in patients who present endometrial compaction at the time of transfer versus those who with a stable or greater endometrial thickness with respect to the estrogenic phase. The estimated duration of the study is 24-30 months. Inclusion criteria are: 18 to 50 years of age, with primary or secondary infertility, subjected to endometrial preparation in a modified natural cycle for transfer of a genetically euploid blastocyst, from their own oocyte or oocyte donation, with a normal uterine cavity. Exclusion criteria are: uterine or endometrial disease (e.g., multiple myomatosis, severe adenomyosis, Asherman syndrome, refractory endometrium), conditions that prevent correct ultrasound assessment (tilted uterus), or a history of recurrent implantation failure or repeated miscarriages.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 50 years
* Primary or secondary infertility
* Normal uterine cavity
* Endometrial preparation in a modified natural cycle for single embryo transfer
* Embryo in blastocyst state from own oocyte or oocyte donation cycles, who had normal results on preimplantation genetic testing for aneuploidy (PGT-A) via trophectoderm biopsy.

Exclusion Criteria:

* Uterine or endometrial disease (multiple myomatosis [>3 fibroids of > 3 cm], adenomyosis, Asherman syndrome)
* Difficulties in correctly measuring endometrial thickness due to a retroverted or tilted uterus
* History of recurrent implantation failure (3 or more transferred blastocysts of good quality, from their own oocyte [<35 years] or oocyte donation); recurrent early Pregnancy Loss (the loss of two or more pregnancies before 10 weeks of gestational age.
* Suboptimal endometrial response (endometrium < 6 mm on the day of ovulation triggering).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women undergoing fertility treatment.
Study Population: 206 Women between 18-50 years, with primary or secondary infertility, undergoing fertility treatment that includes endometrial preparation in a modified natural cycle for transfer of previously analyzed frozen and euploid embryos.
Sampling Method: Non-Probability Sample
Enrollment: 206 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 8-10 weeks gestational age.
  Presence of an intrauterine pregnancy with positive embryo heartbeat as seen by sonography at 8-10 weeks gestational age.

SECONDARY OUTCOMES:
Biochemical pregnancy loss | 9-10 days after the embryo transfer.
  Spontaneous pregnancy demise based on decreasing serum b-hCG levels, without an ultrasound evaluation.
Clinical pregnancy | 5-6 weeks gestational age.
  A pregnancy diagnosed by ultrasonographic visualization of one or more gestational sacs or definitive clinical signs of pregnancy.
Ectopic pregnancy | 5-8 weeks gestational age.
  ultrasonic or surgical visualization of a pregnancy outside of the endometrial cavity.
Early pregnancy loss | 5-10 weeks gestational age.
  spontaneous pregnancy demise before 10 weeks of gestational age (before 8th developmental week).

CONTACTS AND LOCATIONS:
Overall Officials: Juan Carlos J Castillo Farfan, Doctor, Study Director — Instituto Bernabeu Alicante
Locations (1):
- Instituto Bernabeu, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-07-29): https://cdn.clinicaltrials.gov/large-docs/70/NCT05960370/ICF_000.pdf